CLINICAL TRIAL: NCT02252159
Title: Prospective, Non-interventional Study of Disease Progression and Treatment of Patients With Polycythemia Vera in United States Academic or Community Clinical Practices
Brief Title: Prospective Observational Study Of Patients With Polycythemia Vera In US Clinical Practices (REVEAL)
Status: Completed | Type: Observational
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: INCB-MA-PV-401
Record Dates: First submitted 2014-09-23; First posted 2014-09-30 (Estimated); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: MPN (Myeloproliferative Neoplasms)
Keywords: Polycythemia; Polycythemia Vera; Hematologic Diseases; Myeloproliferative Disorders; Bone Marrow Diseases; Hydroxyurea; Antineoplastic Agents; Therapeutic Uses; Pharmacologic Actions; Antisickling Agents; Hematologic Agents; Enzyme Inhibitors; Molecular Mechanisms of Pharmacological Action; Nucleic Acid Synthesis Inhibitors
MeSH Terms: conditions — Myeloproliferative Disorders; Polycythemia; Polycythemia Vera; Hematologic Diseases; Bone Marrow Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample(s), two vials, one with heparin, another with ethylenediaminetetraacetic acid (EDTA) will be collected at enrollment and then annually thereafter until the end of study for serum analysis of proteins and assessment of allele burden and mutations.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort A: Patients with clinically overt PV (and not exhibiting any of the characteristics listed for Cohort B), managed with:
  1. Watchful waiting (with or without aspirin)*, or
  2. Phlebotomy (PHL) alone (with or without aspirin)* - or
  3. HU alone (without concomitant PHL, with or without aspirin).
  (*Unless patient has a history of intolerance or clinical resistance/ refractoriness to hydroxyurea [HU] (as assessed by the treating physician) - in which case, s/he belongs to Cohort B)
- Cohort B: Patients with clinically overt PV, with one or more of the following disease characteristics:
  1. Treatment with HU and PHL in combination or
  2. Treatment with any agent other than HU or aspirin (e.g., recombinant interferon (IFN) or pegylated IFN preparations, busulfan, anagrelide) or
  3. A history of thrombosis (venous or arterial) or
  4. A history of intolerance or clinical resistance/ refractoriness to HU (as assessed by the treating physician) or
  5. Presence of documented splenomegaly (clinically assessed by palpation) or
  6. Presence of one or more of the following uncontrolled symptoms related to PV despite therapy (Symptoms deemed uncontrolled as per physician's judgment)
     1. Tiredness
     2. Difficulty sleeping
     3. Itching
     4. Muscle aches and/or bone pain
     5. Night sweats
     6. Sweats while awake
     7. Other

SUMMARY:
This is a Phase IV, multicenter, non-interventional, non-randomized, prospective, observational study in an adult population (patients >18 years old) of men and women who have been diagnosed with clinically overt PV and are being followed in either community or academic medical centers in the United States who will be enrolled over a 12-month period and observed for 36 months from the date the last patient is enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosis of Polycythemia Vera (PV)
* Willing and able to provide written informed consent
* Willing and able to complete patient assessment questionnaires either alone or with minimal assistance from a caregiver and/or trained site personnel
* Under the supervision of a physician for the current care of PV including but not limited to watchful waiting, acetylsalicylic acid (ASA) 81mg or greater, antithrombotic therapy, Phlebotomy (PHL), Hydroxyurea (HU), interferon (recombinant or pegylated), busulfan, anagrelide

Exclusion Criteria:

* Participation in an active clinical trial in which the study treatment is blinded
* Life expectancy <6 months
* Diagnosis of myelofibrosis (MF) [including primary MF, post-PV MF, or post-essential thrombocythemia MF (post-ET MF)]
* Diagnosis of secondary Acute Myeloid Leukemia (AML)
* Diagnosis of Myelodysplastic Syndrome (MDS)
* History of or active plan to proceed to allogeneic hematopoietic stem cell transplant in next 3 months
* Splenectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: An adult population (patients >18 years old) of men and women who have been diagnosed with clinically overt PV will be enrolled. Sites will include both community and academic centers across the United States that are representative of where patients with PV are diagnosed and treated.
Sampling Method: Probability Sample
Enrollment: 2544 (Actual)
Dates: Start 2014-07-31 (Actual); Primary Completion 2019-08-03 (Actual); Study Completion 2019-08-03 (Actual)

PRIMARY OUTCOMES:
Description of patterns of the disease Polycythemia Vera (PV), and associations of such patterns with patients' exposures or treatments | Every 3 months for approximately 36 months
Incidence (frequency) of disease progression | Every 3 months for approximately 36 months
Incidence (frequency) of healthcare resources utilization | Every 3 months for approximately 36 months
  Healthcare resources were defined as a. Medical visits (including Office visits, ER visits, and hospitalizations), b. phlebotomy (PHL) procedures and c. prescriptions (including PV-related prescriptions, PV-related over-the-counter (OTC) medications, and prescription medications for co-morbid conditions).
Incidence (frequency) of complications due to PV | Every 3 months for approximately 36 months
Incidence (frequency) and description of PV-related symptoms | Every 3 months for approximately 36 months

SECONDARY OUTCOMES:
Incidence (frequency) of adverse events (for those patients on active therapies, including PHL) | Baseline through end of study. Approximately 36 months
Patient-reported outcomes as assessed by Myeloproliferative Neoplasm Symptom Assessment Form Total Symptom Score (MPN-SAF TSS) for assessment of the severity of symptoms | Every 3 months for approximately 36 months
  The MPN-SAF TSS is a validated 10-item instrument that efficiently assesses the prevalence and severity of PV symptoms in both clinical practice and trial settings. Higher scores indicate more severe symptoms and greater inactivity with a possible total score range of 0-100.
Work Productivity and Activity Impairment Questionnaire - Specific Health Problem (WPAI-SHP) score for assessment of work productivity and activity impairment | Every 3 months for approximately 36 months
  WPAI-SHP is a validated 6-item instrument that measures the effect of overall health and specific symptoms on productivity at work and outside of it. All outcomes are presented as a proportion, with 0% representing minimal/no impairment and 100% representing maximal impairment or productivity loss.
European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30) for Health Related Quality of Life (HRQoL) | Every 3 months for approximately 36 months
Caregiver burden | Every 3 months for approximately 36 months
  The amount of health care received by a paid healthcare worker or by an unpaid caregiver
Burden of phlebotomy (PHL) | Every 3 months for approximately 36 months
  A patients self-reported assessment of burden including pain at site, difficulty and inconvenience of scheduling and cost factors.

CONTACTS AND LOCATIONS:
Overall Officials: Robyn M. Scherber, MD, MPH, Study Director — Incyte Corporation
Locations (266):
- United States (264):
  - Green Valley, Arizona
  - Safford, Arizona
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Yuma, Arizona
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - North Little Rock, Arkansas
  - Stuttgart, Arkansas
  - Berkeley, California
  - Burbank, California
  - Corona, California
  - Fountain Valley, California
  - Highland, California
  - Laguna Hills, California
  - Los Alamitos, California
  - Oceanside, California
  - Orange, California
  - Pismo Beach, California
  - Rancho Mirage, California
  - Riverside, California
  - Santa Maria, California
  - Santa Rosa, California
  - Tarzana, California
  - Torrance, California
  - Vallejo, California
  - West Hills, California
  - Whittier, California
  - Aurora, Colorado
  - Colorado Springs, Colorado
  - Fort Collins, Colorado
  - Pueblo, Colorado
  - Middletown, Connecticut
  - Norwich, Connecticut
  - Stamford, Connecticut
  - Washington D.C., District of Columbia
  - Aventura, Florida
  - Boynton Beach, Florida
  - Deerfield Beach, Florida
  - Fort Lauderdale, Florida
  - Hialeah, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Miami Lakes, Florida
  - Ocala, Florida
  - Pembroke Pines, Florida
  - Pensacola, Florida
  - Santa Rosa Beach, Florida
  - Winter Haven, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Austell, Georgia
  - Cartersville, Georgia
  - Columbus, Georgia
  - Douglasville, Georgia
  - Gainesville, Georgia
  - Marietta, Georgia
  - Rome, Georgia
  - Savannah, Georgia
  - Thomasville, Georgia
  - Boise, Idaho
  - Post Falls, Idaho
  - Berwyn, Illinois
  - Chicago, Illinois
  - Danville, Illinois
  - Decatur, Illinois
  - Effingham, Illinois
  - Evanston, Illinois
  - Harvey, Illinois
  - Joliet, Illinois
  - Kewanee, Illinois
  - Macomb, Illinois
  - Maywood, Illinois
  - Morris, Illinois
  - New Lenox, Illinois
  - Normal, Illinois
  - Ottawa, Illinois
  - Park Ridge, Illinois
  - Pekin, Illinois
  - Peoria, Illinois
  - Peru, Illinois
  - Princeton, Illinois
  - Skokie, Illinois
  - Springfield, Illinois
  - Urbana, Illinois
  - Anderson, Indiana
  - Columbus, Indiana
  - Crown Point, Indiana
  - Fort Wayne, Indiana
  - Indianapolis, Indiana
  - Lafayette, Indiana
  - Marion, Indiana
  - Mooresville, Indiana
  - New Albany, Indiana
  - Newburgh, Indiana
  - Terre Haute, Indiana
  - Cedar Rapids, Iowa
  - Iowa City, Iowa
  - Mason City, Iowa
  - Sioux City, Iowa
  - Topeka, Kansas
  - Wichita, Kansas
  - Ashland, Kentucky
  - Danville, Kentucky
  - Hazard, Kentucky
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Mount Sterling, Kentucky
  - Paducah, Kentucky
  - Richmond, Kentucky
  - Alexandria, Louisiana
  - Baton Rouge, Louisiana
  - Marrero, Louisiana
  - Shreveport, Louisiana
  - Rockport, Maine
  - Baltimore, Maryland
  - Bethesda, Maryland
  - Clinton, Maryland
  - Cumberland, Maryland
  - Hagerstown, Maryland
  - Boston, Massachusetts
  - Fairhaven, Massachusetts
  - Lawrence, Massachusetts
  - Pittsfield, Massachusetts
  - Worcester, Massachusetts
  - Ann Arbor, Michigan
  - Battle Creek, Michigan
  - Brighton, Michigan
  - Canton, Michigan
  - Chelsea, Michigan
  - Dearborn, Michigan
  - Detroit, Michigan
  - Flint, Michigan
  - Grand Rapids, Michigan
  - Jackson, Michigan
  - Kalamazoo, Michigan
  - Lansing, Michigan
  - Marquette, Michigan
  - Pontiac, Michigan
  - Saginaw, Michigan
  - Edina, Minnesota
  - Minneapolis, Minnesota
  - Saint Cloud, Minnesota
  - Saint Louis Park, Minnesota
  - Saint Paul, Minnesota
  - Bolivar, Missouri
  - Cape Girardeau, Missouri
  - Kansas City, Missouri
  - St Louis, Missouri
  - Billings, Montana
  - Kalispell, Montana
  - Henderson, Nevada
  - Las Vegas, Nevada
  - Dover, New Hampshire
  - Portsmouth, New Hampshire
  - Brick, New Jersey
  - East Orange, New Jersey
  - Edison, New Jersey
  - Flemington, New Jersey
  - Hackettstown, New Jersey
  - Paramus, New Jersey
  - Somerville, New Jersey
  - Sparta, New Jersey
  - Vineland, New Jersey
  - Farmington, New Mexico
  - Albany, New York
  - Binghamton, New York
  - Brooklyn, New York
  - Cooperstown, New York
  - Corning, New York
  - East Setauket, New York
  - Elmira, New York
  - Herkimer, New York
  - Ithaca, New York
  - Johnson City, New York
  - New York, New York
  - Oneonta, New York
  - Poughkeepsie, New York
  - Rochester, New York
  - Staten Island, New York
  - The Bronx, New York
  - Utica, New York
  - Albemarle, North Carolina
  - Boone, North Carolina
  - Charlotte, North Carolina
  - Clayton, North Carolina
  - Durham, North Carolina
  - Greenville, North Carolina
  - Henderson, North Carolina
  - Hendersonville, North Carolina
  - Hickory, North Carolina
  - Lincolnton, North Carolina
  - Shelby, North Carolina
  - Smithfield, North Carolina
  - Winston-Salem, North Carolina
  - Bismarck, North Dakota
  - Canton, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Dover, Ohio
  - Huber Heights, Ohio
  - Massillon, Ohio
  - Mount Vernon, Ohio
  - Oregon, Ohio
  - Toledo, Ohio
  - West Chester, Ohio
  - Oklahoma City, Oklahoma
  - Beaverton, Oregon
  - Corvallis, Oregon
  - Portland, Oregon
  - Salem, Oregon
  - Allentown, Pennsylvania
  - Bethlehem, Pennsylvania
  - Broomall, Pennsylvania
  - Drexel Hill, Pennsylvania
  - Easton, Pennsylvania
  - Gettysburg, Pennsylvania
  - Hanover, Pennsylvania
  - Hershey, Pennsylvania
  - Kittanning, Pennsylvania
  - Philadelphia, Pennsylvania
  - Quakertown, Pennsylvania
  - Sayre, Pennsylvania
  - Upland, Pennsylvania
  - Wellsboro, Pennsylvania
  - Willow Grove, Pennsylvania
  - York, Pennsylvania
  - Pawtucket, Rhode Island
  - Charleston, South Carolina
  - Hilton Head Island, South Carolina
  - Murrells Inlet, South Carolina
  - Rock Hill, South Carolina
  - Rapid City, South Dakota
  - Sioux Falls, South Dakota
  - Watertown, South Dakota
  - Germantown, Tennessee
  - Jackson, Tennessee
  - Nashville, Tennessee
  - Abilene, Texas
  - Athens, Texas
  - Bryan, Texas
  - Corpus Christi, Texas
  - Galveston, Texas
  - Houston, Texas
  - Jacksonville, Texas
  - Plano, Texas
  - Richardson, Texas
  - Tyler, Texas
  - Ogden, Utah
  - Salt Lake City, Utah
  - Bristol, Virginia
  - Chesapeake, Virginia
  - Falls Church, Virginia
  - Portsmouth, Virginia
  - Suffolk, Virginia
  - Bellingham, Washington
  - Everett, Washington
  - Puyallup, Washington
  - Seattle, Washington
  - Martinsburg, West Virginia
  - Green Bay, Wisconsin
  - Milwaukee, Wisconsin
  - Weston, Wisconsin
- Puerto Rico (2):
  - Bayamón
  - Ponce

REFERENCES:
- [Derived] Gerds AT, Mesa R, Burke JM, Grunwald MR, Stein BL, Squier P, Yu J, Hamer-Maansson JE, Oh ST. Association between elevated white blood cell counts and thrombotic events in polycythemia vera: analysis from REVEAL. Blood. 2024 Apr 18;143(16):1646-1655. doi: 10.1182/blood.2023020232. PMID 38142448
- [Derived] Zwicker JI, Paranagama D, Lessen DS, Colucci PM, Grunwald MR. Hemorrhage in patients with polycythemia vera receiving aspirin with an anticoagulant: a prospective, observational study. Haematologica. 2022 May 1;107(5):1106-1110. doi: 10.3324/haematol.2021.279032. PMID 34162181
- [Derived] Grunwald MR, Burke JM, Kuter DJ, Gerds AT, Stein B, Walshauser MA, Parasuraman S, Colucci P, Paranagama D, Savona MR, Mesa R. Symptom Burden and Blood Counts in Patients With Polycythemia Vera in the United States: An Analysis From the REVEAL Study. Clin Lymphoma Myeloma Leuk. 2019 Sep;19(9):579-584.e1. doi: 10.1016/j.clml.2019.06.001. Epub 2019 Jun 13. PMID 31303457
- [Derived] Mesa R, Boccia RV, Grunwald MR, Oh ST, Colucci P, Paranagama D, Parasuraman S, Stein BL. Patient-Reported Outcomes Data From REVEAL at the Time of Enrollment (Baseline): A Prospective Observational Study of Patients With Polycythemia Vera in the United States. Clin Lymphoma Myeloma Leuk. 2018 Sep;18(9):590-596. doi: 10.1016/j.clml.2018.05.020. Epub 2018 May 28. PMID 30122202
- See also: Related Info — http://www.RevealPVStudy.com